CLINICAL TRIAL: NCT01262352
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Effect of VX-770 on Lung Clearance Index in Subjects With Cystic Fibrosis, the G551D Mutation, and FEV1 >90% Predicted
Brief Title: Study of the Effect of Ivacaftor on Lung Clearance Index in Subjects With Cystic Fibrosis and the G551D Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX10-770-106
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Sequence 1 (Experimental): Ivacaftor administered in Treatment Period 1 and placebo administered in Treatment Period 2.
  Interventions: Drug: Ivacaftor; Drug: Placebo
- Treatment Sequence 2 (Experimental): Placebo administered in Treatment Period 1 and ivacaftor administered in Treatment Sequence 2.
  Interventions: Drug: Ivacaftor; Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor — 150 mg tablet, oral use, twice daily every 12 hours (q12h)
Drug: Placebo — Tablet, oral use, twice daily every 12 hours (q12h)

SUMMARY:
The purpose of this study is to evaluate the effect of ivacaftor (VX-770) on lung clearance index (LCI) in subjects aged 6 years and older with cystic fibrosis (CF) who have the G551D-CFTR mutation on at least 1 allele.

DETAILED DESCRIPTION:
Currently, limited objective measures are available to quantify lung function in CF patients with mild lung disease. Lung clearance index (LCI) derived from inert gas multiple-breath washout (MBW) testing hold considerable promise to evaluate early lung disease as studies have detected abnormalities in a high percentage of CF patients with normal spirometry in both infants and children.

This study explored the effect of ivacaftor on LCI and the efficacy of ivacaftor on other clinical and biomarker endpoints of CF lung disease in subjects aged 6 years and older with CF who have the G551D-CFTR mutation on at least 1 allele.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with confirmed diagnosis of CF
* Must have the G551D-CFTR mutation in at least 1 allele
* FEV1 >90% of predicted normal for age, gender, and height

Exclusion Criteria:

* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within the 30 days prior to screening
* Use of inhaled hypertonic saline treatment within 2 weeks of the Period 1, Day 1 visit

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Davies, Principal Investigator — Royal Brompton Hospital and Imperial College; Felix Ratjen, Principal Investigator — The Hospital for Sick Children
Locations (8):
- United States (4):
  - Stanford, California
  - Iowa City, Iowa
  - Durham, North Carolina
  - Pittsburgh, Pennsylvania
- Toronto, Ontario, Canada
- United Kingdom (3):
  - Belfast
  - Edinburgh
  - London

REFERENCES:
- [Derived] Davies J, Sheridan H, Bell N, Cunningham S, Davis SD, Elborn JS, Milla CE, Starner TD, Weiner DJ, Lee PS, Ratjen F. Assessment of clinical response to ivacaftor with lung clearance index in cystic fibrosis patients with a G551D-CFTR mutation and preserved spirometry: a randomised controlled trial. Lancet Respir Med. 2013 Oct;1(8):630-638. doi: 10.1016/S2213-2600(13)70182-6. Epub 2013 Sep 10. PMID 24461666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started on 14 February 2011 (signing of first informed consent). After obtaining informed consent and assent (where applicable), screening evaluations were completed at any time during the period 10 to 18 days (Days -18 to -10) before first dose of study drug (Day 1).
Pre-assignment Details: A total of 21 subjects were randomized; 20 subjects received at least 1 dose of the study drug.
Groups:
- Ivacaftor Then Placebo: Ivacaftor administered in Treatment Period 1 and placebo administered in Treatment Period 2.
- Placebo Then Ivacaftor: Placebo administered in Treatment Period 1 and ivacaftor administered in Treatment Period 2.
Period: Period 1
Arm/Group | Ivacaftor Then Placebo | Placebo Then Ivacaftor
Started | 11 | 10
Dosed | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Illness after randomization | 1 | 0
Period: Washout
Arm/Group | Ivacaftor Then Placebo | Placebo Then Ivacaftor
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Extended Washout | 0 | 1
Period: Period 2
Arm/Group | Ivacaftor Then Placebo | Placebo Then Ivacaftor
Started | 9 | 8
Dosed | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivacaftor Then Placebo | Placebo Then Ivacaftor | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 7 | 16
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.4 (7.12) | 19.8 (13.35) | 16.6 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 6 | 5 | 11
  Europe | 4 | 5 | 9
Height [Mean (Standard Deviation); unit: centimeters] | 148.9 (19.54) | 156.0 (17.92) | 152.5 (18.61)
Weight [Mean (Standard Deviation); unit: kilograms] | 45.06 (20.018) | 58.78 (30.576) | 51.92 (26.119)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 19.36 (3.707) | 22.66 (6.964) | 21.01 (5.687)
Lung Clearance Index (LCI) [Mean (Standard Deviation); unit: ratio] — Lung clearance index (LCI) is a measure of ventilation inhomogeneity that is derived from a multiple-breath washout test. The LCI was calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity [FRC]) required to reduce end-tidal SF6 concentration to 1/40th of the starting value.
  ratio | 9.17 (1.657) | 8.88 (1.462) | 9.03 (1.528)
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percentage] | 101.83 (11.587) | 92.58 (7.427) | 97.20 (10.595)
Sweat Chloride [Mean (Standard Deviation); unit: millimoles per liter] | 97.10 (7.400) | 86.17 (19.219) | 91.92 (14.933)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Lung Clearance Index (LCI)
Description: Lung clearance index (LCI) is a measure of ventilation inhomogeneity that is derived from a multiple-breath washout test. The LCI was calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity [FRC]) required to reduce end-tidal SF6 concentration to 1/40th of the starting value.
Time Frame: Baseline through Day 29
Population: All randomized subjects who received at least 1 dose of study drug (placebo or ivacaftor) and had available assessments during the time frame.
Measure: Least Squares Mean (Standard Error); unit: ratio
Groups:
- Placebo: Oral tablet every 12 hours (q12h) for up to 28 days.
- Ivacaftor: Oral tablet of 150 mg of ivacaftor q12h for up to 28 days.
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 18 | 17
ratio | 0.77 (0.291) | -1.30 (0.303)
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; The primary analysis for the primary efficacy variable was based on a mixed effect model. The model included the absolute change from the baseline in each period as the dependent variable, sequence, treatment, and period as fixed effects, study baseline LCI as the covariate, and subject nested within sequence as the random effect; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -2.069, 95% CI 2-sided [-2.98 to -1.15]

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted FEV1
Description: Spirometry (as measured by FEV1) is a standardized assessment to evaluate lung function that is the most widely used endpoint in cystic fibrosis studies.
Time Frame: Baseline through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 19 | 18
percent | 0.00 (1.916) | 7.00 (1.978)
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Analysis for this efficacy variable was performed in a similar way as the analysis for the primary efficacy variable; Test type: Superiority or Other; p = 0.0117, Mixed Models Analysis — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 7.007, 95% CI 2-sided [1.80 to 12.21]

3. Secondary Outcome: Change From Baseline in Sweat Chloride
Description: The sweat chloride (quantitative pilocarpine iontophoresis) test is a standard diagnostic tool for cystic fibrosis (CF), serving as an indicator of cystic fibrosis transmembrane conductance regulator (CFTR) activity.
Time Frame: Baseline through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 18 | 16
millimoles per liter | 0.11 (2.351) | -45.74 (2.632)
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; Analysis for change from baseline in average sweat chloride was similar to the analysis of the primary efficacy variable; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -45.848, 95% CI 2-sided [-53.54 to -38.16]

4. Secondary Outcome: Change From Baseline in CF Questionnaire-Revised (CFQ-R) Score (Respiratory Domain Score, Pooled)
Description: The CFQ-R is a health-related quality of life measure for subjects with cystic fibrosis. Each domain is scored from 0 (worst) to 100 (best). A difference of at least 4 points in the respiratory domain score of the CFQ-R is considered a minimal clinically important difference (MCID). The primary analytical focus was the respiratory health domain, which was analyzed by combining all self-response questionnaire versions from different age groups (e.g., Adult/Adolescent and Child versions).
Time Frame: Baseline through Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ivacaftor
Number analyzed (Participants) | 19 | 18
score on a scale | 1.33 (3.067) | 5.32 (3.166)
Statistical Analysis 1: Comparison: Placebo vs Ivacaftor; The raw scores in CFQ-R were summarized into different domains of health (12 domains for adolescents and adults 14 years of age and older, 8 domains for children ages 12 and 13 years, 8 domains for children ages 6 to 11 years, and 11 domains for parents/caregivers). Each domain was analyzed in a similar way as for the primary efficacy variable. The primary analytical focus was the respiratory health domain which was analyzed by combining all self-response questionnaire versions; Test type: Superiority or Other; p = 0.3796, Mixed Models Analysis — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 3.991, 95% CI 2-sided [-5.40 to 13.39]

ADVERSE EVENTS:
Time Frame: For enrolled subjects, all adverse events were collected through the Follow-up Visit (4 weeks [+/-7 days] after the last dose of study drug).
Description: For subjects who were screened but were not subsequently enrolled in the study, all adverse events were collected until the subject was deemed ineligible for the study.
Arm/Group | Placebo | Ivacaftor
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/18
Other Adverse Events (participants affected / at risk) | 15/19 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Ivacaftor (N=18)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Ivacaftor (N=18)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Application site papules (General disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Mycobacterium abscessus infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bacteria sputum identified (Investigations) | 0 (0) | 1 (1)
Bacterial culture positive (Investigations) | 1 (1) | 0 (0)
Lymph node palpable (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.